CLINICAL TRIAL: NCT05325398
Title: Effect of Molecular Hydrogen in Patients With Non Alcoholic Faty Liver Disease
Brief Title: Effect of Molecular Hydrogen in Patients With NAFLD
Acronym: EMoHyNAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Collaborators: NWN & Drink HRW (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/2020/UNB/IIIrdInternal
Record Dates: First submitted 2021-05-14; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Molecular hydrogen; effective antioxidant; oxygen radicals; NAFLD; mitochondria
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with NAFLD (Active Comparator): 17 patients will receive molecular hydrogen
  Interventions: Dietary Supplement: HRW drink, HRW Natural Health Products Inc., Made in Vancouver, Canada
- probands in the control group (Placebo Comparator): 13 probands in the control group who will receive placebo.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: HRW drink, HRW Natural Health Products Inc., Made in Vancouver, Canada — The cohort will consist of 17 patients with NAFLD. Name of the product that will be the source of molecular hydrogen: HRW drink, HRW Natural Health Products Inc., Made in Vancouver, Canada. It is a nutritional supplement that is a source of molecular hydrogen.
  All study participants will drink one tablet dissolved in 0.33 l of tap water every 8 hours.
  They did this for 8 weeks. Blood analysis at study entry and after 8 weeks (end of study).
  Arms: patients with NAFLD
Dietary Supplement: placebo — 13 probands in the control group who will receive placebo. All study participants will drink one placebo tablet dissolved in 0.33 l of tap water every 8 hours.
  They did this for 8 weeks. Blood analysis at study entry and after 8 weeks (end of study)
  Arms: probands in the control group

SUMMARY:
Molecular hydrogen H2 acts as antioxidant which selectively reduces cytotoxic harmful reactive oxygen species ROS and concomitantly acts as biological messenger, which mediates several signaling pathways that play cytoprotective role in many human diseases. Due to their small size and high permeability, H2 is easily transportable into subcellular structures as mitochondria.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease, NAFLD, is the most common cause of liver disease. According to the forecasts, the non-alcoholic steatohepatitis will be the most common cause of liver transplantation and hepatic mortality in 2030. NAFLD is also a significant risk factor for the development of hepatocellular carcinoma, even in the non-cirrhotic stage of liver disease. The prevention of the progression of NAFLD to NASH (nonalcoholic steatohepatitis) is therefore a key factor in preventing this unfavorable prognosis.

Obesity and its associated comorbidities are among the most widespread and challenging conditions in the confrontation of the medical profession in the 21st century. The main metabolic consequence of obesity is insulin resistance, which is strongly associated with the storage of triacylglycerols in the liver. Hepatic steatosis may be associated with steatohepatitis, a condition that can lead to liver cirrhosis and, in the final stage, liver transplantation.

According to various sources, the incidence of NAFLD in the population is 20-30%, in obese up to 60%, which makes it the most common liver disease. In the USA, it is even 3 times more common than type 2 diabetes mellitus and 5-10 times more common than chronic hepatitis C. The incidence of non-alcoholic steatohepatitis NASH is 2-3% and is now thought to be the cause of up to 80% cryptogenic liver cirrhosis. The risk of developing cirrhosis in patients with simple hepatic steatosis is 1-2% over 8 years.

Insulin resistance, which is defined as an elevated HOMA (homeostasis model assessment) index above 1,4, is found in 70% of patients with NAFLD and plays a major role in the accumulation of triacylglycerols TAG (triacylglyceride) in the liver. Through the rise of hormone-sensitive lipase, hyperinsulinemia leads to the hydrolysis of free fatty acids FFA from visceral adipocytes to the portal vein, through which they enter directly into the liver, where they are esterified to TAG. Reducing the production of apolipoprotein B-100, which is an important part of their secretion from the liver into the circulation in the form of VLDL-lipoproteins, is also a potentiating factor in TAG deposition in the liver. Free oxygen radicals ROS (reactive oxygen species), which are formed due to the oxidative stress, are formed directly in the hepatocyte. However, their formation in visceral adipocytes has also been shown to be involved in liver damage. The main site of ROS are mitochondria. In NAFLD, known mitochondrial dysfunction leads to pathological oxidation of FFA (free fatty acid) in peroxisomes and microsomes, making them another source of ROS. ROS, through damage of the mitochondrial membrane by lipoperoxidation and induction of Fas-ligand expression on the hepatocyte, leads to cell apoptosis.

By activating stellate cells, a larger amount of extracellular matrix is formed - Mallory's hyaline, which is associated with the formation of balloon degeneration of hepatocytes, that is a typical histological feature of NASH.

From the cytokines, TNF-alpha is mainly used. It is formed by hepatocytes due to the increased supply of FFA. The diagnostic process is often random. One of the options for non-invasive measurement of liver fibrosis is transient elastography FibroScan, which is used for direct measurement of liver elasticity or use of noninvasive fibrosis indexes (NFS, Fib-4, APRI etc) as nondirect tools. Initial studies have confirmed that H2 penetrates cell membranes and protects mitochondria and cell nuclei from acute oxidative stress. Several studies have reported the effect of H2 on mitochondrial function. With H2, the investigators protect the potential of the mitochondrial membrane, increase ATP production and reduce organelle swelling. There are at least four possible mechanisms for H2 through which gene expression can be altered through mitochondrial bioenergetics, of which ghrelin is probably the most important. Ghrelin is the hormone responsible for appetite.

It reaches its maximum level during hunger. Obestatin has the opposite effect, which in turn suppresses the feeling of hunger. The role of ghrelin as an energy modulator in H2 intervention may be promoted by interaction with expressed glucose transporters, which increase glucose consumption and modulate oxidative phosphorylation in mitochondria. Exercise led to a significant change in ghrelin levels but had no effect on plasma levels of obestatin.

Molecular hydrogen has been shown to relieve oxidative stress, have an anti-inflammatory effect and improve lipid, glucose and energy production in patients as well as in animal models of hepatic steatosis and atherosclerosis. The basic molecular mechanisms remain largely unknown.

Molecular hydrogen is an effective antioxidant that reduces cytotoxic reactive oxygen radicals, especially the hydroxyl radical. In several previous experiments, the use of hydrogen-enriched water, HRW, has been shown to have antioxidant effects. The effects of hydrogen on the prevention of hepatocarcinogenesis in STAM mice were also investigated. The number of tumors was significantly lower in the HRW groups and the tumors were smaller than in the other groups. The results clearly demonstrated that HRW can be an effective treatment for apoptosis, inflammation and hepatocarcinogenesis in NAFLD.

The aim of the study is to verify effectiveness and safety of molecular hydrogen on a group of patients with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* People with age 33-69 years
* BMI ≥ 25
* Confirmation of fatty liver by ultrasonographic examination
* Signed informed consent
* Alcohol intake according to the AUDIT questionnaire 5 or less points for men or 4 or less points for women

Exclusion Criteria:

* Unsigned informed consent
* BMI < 25
* Presence of severe inflammatory disease with activity (Crohn's disease, ulcerative colitis, active tuberculosis, rheumatoid arthritis, etc.)
* Presence of acute infectious disease (acute hepatitis, peritonitis, cholecystitis, pancreatitis, etc.)
* Presence of active neoplastic disease
* Alcohol intake according to the AUDIT questionnaire more as 5 points for men or more as 4 points for women

Ages: 33 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Changes in body parameters: Weight in kilograms, height in meters, waist circumference in centimeters | 8 weeks
  The following parameters will be measured for each proband before (time 0) and after the study (time 8 weeks):
  a) weight and height will be combined to report BMI in kg/m^2, waist circumference in cm.
Changes in blood parameters ALT | 8 weeks
  ALT (alaninaminotransferase) ukat/L
Changes in blood parameters AST | 8 weeks
  AST (aspartataminotransferase) ukat/L
Changes in blood parameters ALP | 8 weeks
  ALP (alkaline phosphatase) ukat/L
Changes in blood parameters GMT | 8 weeks
  GMT (gamaglutamyltransferase) ukat/L
Changes in blood parameters Albumin | 8 weeks
  Albumin (g/L)
Changes in blood parameters Cholinesterase | 8 weeks
  Cholinesterase (ukat/L)
Changes in blood parameters Bilirubin | 8 weeks
  Bilirubin total (umol/L)
Changes in blood parameters Glucose | 8 weeks
  Glucose (mmol/L)
Changes in blood parameters Cholesterol | 8 weeks
  Cholesterol (mmol/L)
Changes in blood parameters Triacylglycerol | 8 weeks
  Triacylglycerol (mmol/L)
Changes in blood parameters Insulin | 8 weeks
  Insulin (mIU/L)
Changes in blood parameters HOMA index | 8 weeks
  HOMA index (calculation)
Changes in blood parameters Leucocytes | 8 weeks
  Leucocytes (x10^9/L)
Changes in blood parameters Hemoglobin | 8 weeks
  Hemoglobin (g/L)
Changes in blood parameters Platelets | 8 weeks
  Platelets (x10^9/L)
Changes in blood parameters TBARS | 8 weeks
  TBARS (μmol/L)
Changes in blood parameters MDA | 8 weeks
  MDA (malondialdehyde) (μmol/L)
Changes in blood parameters LDH | 8 weeks
  LDH (lactatdehydrogenase) (mU/mL)
Changes in blood parameters MMP-2 | 8 weeks
  MMP-2 (matrix metalloproteinase2) (% of change)
Changes in blood parameters MMP-9 | 8 weeks
  MMP-9 (matrix-metalloproteinase 9) (% of change)
Changes in blood parameters 8-OHdG | 8 weeks
  8-OHdG (8-hydroxy-2-deoxyguanosine) (ng/mL)
Changes in blood parameters SOD | 8 weeks
  SOD (superoxiddismutase) (ng/mL)
Changes in blood parameters NFkB | 8 weeks
  NFkB (nuclear factor kappa B) (% of change)
Changes in blood parameters TNF alfa | 8 weeks
  TNF alfa (tumor necrosis factor alpha) (% of change)
Changes in blood parameters HSP 60 | 8 weeks
  HSP 60 (heat shock protein 60) (% of change)
Changes in blood parameters HSP 70 | 8 weeks
  HSP 70 (heat shock protein 70) (% of change)
Changes in blood parameters Alpha tocopherol | 8 weeks
  Alpha tocopherol (μmol/L)
Changes in blood parameters Gama tocopherol | 8 weeks
  Gama tocopherol (μmol/L)
Changes in blood parameters Beta carotene | 8 weeks
  Beta carotene (μmol/L)
Changes in blood parameters Coenzyme Q 10 in platelets | 8 weeks
  Coenzyme Q 10 in platelets (pmol/10^9 cells)
Changes in blood parameters Coenzyme Q 10 in plasma | 8 weeks
  Coenzyme Q 10 in plasma (μmol/L)
Changes in blood parameters Coenzyme Q 10 in whole blood | 8 weeks
  Coenzyme Q 10 in whole blood (μmol/L)

OTHER OUTCOMES:
Entry check of patients health status- clinical examination SPG and SPL | 2 hours
  Entry examination will include:
  SPG: Status presens generalis (consciousness, body habitus, skin, nutrition), SPL: status presens localis (head, neck, chest, abdomen, limbs)- described generally as number of participants with changes in healt status
Entry check of patients health status- urinary sediment | 2 hours
  Urinary sediment normal : leucocyte 1-2 , erythrocyte: 0-1, cultivation: negative or bacterial agens more than 10^5 - described generally as number of participants with changes in urinary sedinent status (normal/abnormal)
Entry check of patients health status- USG | 2 hours
  USG: Ultrasonographic examination: fatty liver: enlargement of the liver more than 130 mm in anteroposterior position, enlarged echogenity of the liver, curved anterior liver lobe. 1 of these parameter is sufficient for diagnosis of fatty liver - described generally as number of participants with changes in urinary sedinent status (normal/abnormal)
Entry check of patients health status- Life style risk factors questionnaire | 1 hours
  Filling of the following Questionnaire: Life style risk factors questionnaire Part A/ NAFLD score more as 7 points means risk of nonalcoholic fatty liver disease (NAFLD) Minimum: 0 points Maximum: 14 points Part. B/ ALD score (AUDIT C questionnaire) more than 5 points = risk of alcoholic liver disease (ALD) Minimum: 0 points Maximum: 12 points 5 points and more = risk of ALD , risk of worse outcome
Entry check of patients health status- AUDIT questionnaire of alcohol intake | 30 minutes
  Filling of the following Questionnaire: AUDIT questionnaire of alcohol intake Minimum: 0 points Maximum: 40 points 8 points and more= risky alcohol drinking , risk of ALD , risk of worse outcome
Entry check of patients health status- Fast Depression screening by Patient Health Questionnaire | 10 minutes
  Filling of the following Questionnaire: Fast Depression screening by Patient Health Questionnaire (2 questions) Minimum: 0 points Maximum: 6 points 3 points and more: risk for depression, risk of worse outcome
Entry check of patients health status- Generalized Anxiety Disorder | 10 minutes
  Filling of the following Questionnaire: Generalized Anxiety Disorder (2 questions) Minimum: 0 points Maximum: 4 points 3 points and more: risk for generalized anxiety disorder, risk of worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- 3rd Department of Internal Medicine Faculty of Medicine Comenius University in Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gvozdjakova A, Klauco F, Kucharska J, Sumbalova Z. Is mitochondrial bioenergetics and coenzyme Q10 the target of a virus causing COVID-19? Bratisl Lek Listy. 2020;121(11):775-778. doi: 10.4149/BLL_2020_126. PMID 33164536
- [Background] Gvozdjakova A, Sumbalova Z, Kucharska J, Komlosi M, Rausova Z, Vancova O, Szamosova M, Mojto V. Platelet Mitochondrial Respiration, Endogenous Coenzyme Q10 and Oxidative Stress in Patients with Chronic Kidney Disease. Diagnostics (Basel). 2020 Mar 23;10(3):176. doi: 10.3390/diagnostics10030176. PMID 32210203
- [Background] Gvozdjakova A, Kucharska J, Sumbalova Z, Rausova Z, Chladekova A, Komlosi M, Szamosova M, Mojto V. The importance of coenzyme Q10 and its ratio to cholesterol in the progress of chronic kidney diseases linked to non- -communicable diseases. Bratisl Lek Listy. 2020;121(10):693-699. doi: 10.4149/BLL_2020_113. PMID 32955899
- [Background] Gvozdjakova A, Kucharska J, Sumbalova Z, Nemec M, Chladekova A, Vancova O, Rausova Z, Kubalova M, Kuzmiakova Z, Mojto V. Platelets mitochondrial function depends on CoQ10 concentration in winter, not in spring season. Gen Physiol Biophys. 2019 Jul;38(4):325-334. doi: 10.4149/gpb_2019012. Epub 2019 Jun 26. PMID 31241044
- [Background] Gvozdjakova A, Sumbalova Z, Kucharska J, Chladekova A, Rausova Z, Vancova O, Komlosi M, Ulicna O, Mojto V. Platelet mitochondrial bioenergetic analysis in patients with nephropathies and non-communicable diseases: a new method. Bratisl Lek Listy. 2019;120(9):630-635. doi: 10.4149/BLL_2019_104. PMID 31475544